CLINICAL TRIAL: NCT04250870
Title: COMPARISON OF THE PHYSICAL FITNESS LEVELS IN NURSING HOME RESIDENTS AND COMMUNITY DWELLING ELDERLY PEOPLE
Brief Title: Physical Fitness in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Yuruk, PT, PHD, Assoc Prof, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KA18/434
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Aging; Healthy Aging; Physical Fitness
Keywords: aging; community dwelling; health; nursing homes; physical fitness

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing Home Residents (Active Comparator): Nursing home residents (n=59) were evaluated in five different nursing homes.
  Interventions: Diagnostic Test: Senior Fitness Test
- Community-Dwelling Elderly (Active Comparator): The community-dwelling elderly people (n=59) were selected from two different municipalities of the city.
  Interventions: Diagnostic Test: Senior Fitness Test

INTERVENTIONS:
Diagnostic Test: Senior Fitness Test — Chair stand test:The number of full stands performed on a seated position that can be completed within 30 seconds was recorded.
  Arm curl test: The participants were asked to lift weights starting with a full elbow extension and then full flexion.
  2-minute step test: The participant was asked to begin stepping as quickly as possible to reach the marked height for two minutes.
  Chair sit-and-reach test:The participant could extend right or left knee to a full extension, heel on the floor and ankle in a neutral position of 90 degrees. Then, the participant was asked to reach to the toes.
  Back-scratch test:The participant was asked to stand up and place his/her preferred hand over the same shoulder, palm down and fingers extended, and reach down the middle of the back as far as possible.
  8-foot up and go test:The participant was asked to get up from a chair without any arm support and walk a distance of 2.44 meters; then turn around a cone and come back to sit down on the chair.

SUMMARY:
Aging decreases the physical fitness levels in living beings. The environmental factors also have a major effect on the physical fitness levels. The objective of this study was to compare the physical fitness levels of nursing home residents and community-dwelling elderly people. This study employed 118 participants, who consisted of nursing home residents and community-dwelling elderly people. The physical fitness levels of the elderly people were measured by Senior Fitness Test. The physical fitness levels of the elderly people were measured by Senior Fitness Test. Chair stand test, arm curl test, 2-minute step test, chair sit and reach test, back-scratch test, 8-foot up and go test and body mass index were measured.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 65 and 85 years
2. Scored between 24 and 30 points in the Mini-Mental Status Examination (MMSE).
3. Living in nursing homes for at least six months (for nursing home residents) (6,7).

Exclusion Criteria:

1. Not able to communicate verbally
2. Not able to stand for at least 90 seconds and ambulated with assistance
3. Patients with severe visual impairment, neurological disorders and/or congestive heart failure
4. Individuals who are not advised exercise.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
2-minute step test | 2 hours
  The distance from the iliac crest to the midpoint of the patella was measured by a tape to determine the knee-stepping height. The midpoint of the distance between these two anatomical structures was determined. The height of the determined point from the ground was measured and marked on the wall. The participant was asked to begin stepping as quickly as possible to reach the marked height for two minutes. The total number of correct dominant side steps was recorded. If any of the participant's steps (right or left) did not reach the target height, those steps were considered invalid.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No